CLINICAL TRIAL: NCT04076722
Title: Neurotrophic Indicators of Cognition, Executive Skills, Plasticity, and Adverse Childhood Experiences Study "NICE SPACES"
Brief Title: Neurotrophic Indicators of Cognition, Executive Skills, Plasticity, and Adverse Childhood Experiences Study
Acronym: NICE SPACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: AS1965
Record Dates: First submitted 2019-07-24; First posted 2019-09-03 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Weight Loss; Wait-List Control
Keywords: Obesity; Weight Loss; Adverse childhood experiences; Executive function; Brain health
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study condition (weight stigma vs. not stigma) was contained in a blinded envelope that only the confederate had access to. The PI does not know which condition the participant got. And the outcomes assessors did not know the condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress reactivity weight stigma (Experimental): This study arm received a stress reactivity paradigm that involved weight stigma content in the form of an evaluated speech task.
  Interventions: Behavioral: Stress reactivity stimuli
- Stress reactivity non-weight stigma. (Active Comparator): This study arm received a stress reactivity paradigm that involved non-weight stigma content in the form of an evaluated speech task.
  Interventions: Behavioral: Stress reactivity stimuli

INTERVENTIONS:
Behavioral: Stress reactivity stimuli — An evaluated speech task delivered to participants after baseline testing.

SUMMARY:
Adverse childhood experiences (ACEs) are repeatedly shown to predict negative biopsychosocial health outcomes, including obesity. High rates of ACEs in communities are often paralleled by high obesity rates, and higher ACEs, such as child abuse, have been shown to positively predict later obesity and use of unhealthy weight control behaviors. Thus, in light of the high prevalence of and potential causal links between early-life stress and obesity, there is a critical need to further explore the ACEs-obesity relationship in order to understand and to improve obesity outcomes. Given the adverse impact of ACEs and obesity on brain health, two potential high impact treatment targets of the ACEs-obesity relationship will be explored in the proposed pilot study: 1) markers of neurocognition (i.e., executive function; EF) and, 2) brain health/plasticity (i.e., neurotrophins like brain-derived neurotropic factor; BDNF and glial cell derived neurotrophic factor; GDNF).

Specifically, this trial will be the first to 1) Identify whether brain markers of neural health (e.g., neurotrophins) are related to ACES and/or neurocognitive EF performance, and 2) Test whether neuronal or glial neurotrophins predict or change in response to weight loss. Addressing these two needs advances the science of whether ACEs and EF levels are differentially related to brain indices of neural and glial health/plasticity. Results of this pilot may identify a neural substrate and/or profile by which ACEs promote obesity that may ultimately be more amenable to pharmacologic intervention in order to promote weight loss outcomes.

This group-treatment trial will assess 48 obese adults randomized to either an 8-week behavioral weight loss treatment group (n=24) or a wait list control (n=24). Our primary endpoints are percent reductions in body weight and changes in neurotrophins (e.g., BDNF, GDNF). Weight and blood specimens will be assessed at baseline, post-treatment (8-weeks), and follow-up (12-weeks). In testing these endpoints, we will meet the following aims: 1) To test whether neurotrophins are related to ACEs and executive function (EF), and 2) To test if neurotrophins predict or change in response to weight loss trajectory.

****The above description describes the study design that was terminated prematurely due to Covid-19. The following description is the modified protocol.

The treatment described above was canceled and the present study focused on the baseline visit. In this visit, participants participated in a stress reactivity protocol, so instead of looking at change in BDNF, GDNF, and inflammatory markers after weight loss treatment, we looked at change in BDNF, GDNF, and inflammatory markers after the stress activity task. This information will tell us about how ACEs status is related to these biomarkers at baseline and in response to stress.

DETAILED DESCRIPTION:
Adverse childhood experiences (ACEs) are repeatedly shown to predict negative biopsychosocial health outcomes, including obesity. High rates of ACEs in communities are often paralleled by high obesity rates, and higher ACEs, such as child abuse, have been shown to positively predict later obesity and use of unhealthy weight control behaviors. Thus, in light of the high prevalence of and potential causal links between early-life stress and obesity, there is a critical need to further explore the ACEs-obesity relationship in order to understand and to improve obesity outcomes. Given the adverse impact of ACEs and obesity on brain health, two potential high impact treatment targets of the ACEs-obesity relationship will be explored in the proposed pilot study: 1) markers of neurocognition (i.e., executive function; EF) and, 2) brain health/plasticity (i.e., neurotrophins like brain-derived neurotropic factor; BDNF and glial cell derived neurotrophic factor; GDNF).

Specifically, this trial will be the first to 1) Identify whether brain markers of neural health (e.g., neurotrophins) are related to ACES and/or neurocognitive EF performance, and 2) Test whether neuronal or glial neurotrophins predict or change in response to weight loss. Addressing these two needs advances the science of whether ACEs and EF levels are differentially related to brain indices of neural and glial health/plasticity. Results of this pilot may identify a neural substrate and/or profile by which ACEs promotes obesity that may ultimately be more amenable to pharmacologic intervention in order to promote weight loss outcomes.

This group-treatment trial will assess 48 obese adults randomized to either an 8-week behavioral weight loss treatment group (n=24) or a wait list control (n=24). Our primary endpoints are percent reductions in body weight and changes in neurotrophins (e.g., BDNF, GDNF). Weight and blood specimens will be assessed at baseline, post-treatment (8-weeks), and follow-up (12-weeks). In testing these endpoints, we will meet the following aims: Aim 1 - To test whether neurotrophins are related to ACEs and executive function (EF), and Aim 2: To test if neurotrophins predict or change in response to weight loss trajectory. To ensure the success of the trial, we have assembled a team of experts in adult behavioral obesity treatment (PI: Hawkins, PhD), neurotrophins (Consultant: Vasquez, PhD), and biostatistics (Consultant: Washburn, PhD). The results of this study will advance the science of neurocognitive risk of weight loss difficulties and their potential treatment. Our approach ensures that the neurocognitive testing and weight loss protocol can be delivered by trained non-experts, improving its scalability and future dissemination potential. The results could ultimately be used to tailor weight loss treatments such that neurocognitive risk factors related to ACES are identified early and may ultimately be proactively mitigated early in treatment to maximize participants' lasting weight loss outcomes.

****The above description describes the study design that was terminated prematurely due to Covid-19. The following description is the modified protocol.

The treatment described above was canceled and the present study focused on the baseline visit. In this visit, participants participated in a stress reactivity protocol, so instead of looking at change in BDNF, GDNF, and inflammatory markers after weight loss treatment, we looked at change in BDNF, GDNF, and inflammatory markers after the stress activity task. This information will tell us about how ACEs status is related to these biomarkers at baseline and in response to stress.

ELIGIBILITY:
Inclusion Criteria:

* an overweight/obese body mass index (BMI = 25 kg/m2 or greater)
* English speaking
* No use of weight loss medications in the past 3 months,
* No history of or planning to undergo bariatric surgery during the study period,
* Not currently pregnant or breastfeeding or planning to become pregnant during the study period,
* Not already enrolled in a weight loss program (e.g., Weight Watchers ®),
* No significant medical or psychiatric comorbidities, including uncontrolled metabolic disorders (e.g., thyroid, renal, liver), diabetes, heart disease, stroke, cancer, eating disorder, psychosis, mania, dementia, etc.,
* Physician determination that the study is appropriate or safe,
* Able to comply with the assessment procedures
* Able to provide informed consent or assent,
* Not planning to move during study period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals must be biologically female to be eligible for the study.
Enrollment: 55 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Neurotrophins - Brain-Derived Neurotrophic Factor (BDNF) | Baseline (time 0; pre-stressor), Post-stressor (time 1; 30 minutes), Post-stressor (time 2; 60 minutes), Post-stressor (time 3; 90 minutes), ,
  Changes in BDNF
Neurotrophins - Glial-Derived Neurotrophic Factor (GDNF) | Baseline (time 0; pre-stressor), Post-stressor (time 1; 30 minutes), Post-stressor (time 2; 60 minutes), Post-stressor (time 3; 90 minutes), ,
  Changes in GDNF

SECONDARY OUTCOMES:
Inflammatory Panel - IL-6, IL-1beta, TNF-alpha, IFN-gamma | Baseline (time 0; pre-stressor), Post-stressor (time 1; 30 minutes), Post-stressor (time 2; 60 minutes), Post-stressor (time 3; 90 minutes), ,
  Changes in pro-inflammatory cytokines IL-6, IL-1beta, TNF-alpha, INF-gamma

CONTACTS AND LOCATIONS:
Overall Officials: Misty Hawkins, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States